CLINICAL TRIAL: NCT03021551
Title: Oxygen Reserve Index: Utility as Early Warning for Desaturation in Morbidly Obese Patients
Status: Completed | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FLEM0004
Record Dates: First submitted 2017-01-11; First posted 2017-01-16 (Estimated); Results first posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Morbid Obesity; Surgery
Keywords: oxygen; desaturation; obesity
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Rainbow sensor (Experimental)
  Interventions: Device: Rainbow sensor

INTERVENTIONS:
Device: Rainbow sensor — Masimo Radical-7 and Root System with ORi parameter in all subjects are enrolled in the test group and receive an Rainbow sensor during their elective surgery.

SUMMARY:
The Oxygen Reserve Index (ORi) is a reference that could help clinicians with their assessments of normoxic and hyperoxic states by scaling the measured absorption information between 0.00 and 1.00. An ORi of 0.00 corresponds to partial pressure of oxygen (PaO2) values of 100 mmHg and below and an ORi of 1.00 corresponds to PaO2 values of 200 mmHg and above. This is clinical study designed to evaluate the clinical utility of the Oxygen Reserve Index (ORI) as an early warning for arterial hemoglobin desaturation during the induction of general anesthesia and tracheal intubation in obese patients undergoing elective surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* BMI>30, <40 m/kg2
* Control group only: BMI >18.5 m/kg2, <25 m/kg2
* Scheduled for an elective surgical procedure requiring general anesthesia and endotracheal intubation

Exclusion Criteria

* Age less than 18 years
* Adults unable to give primary consent
* Pregnancy
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah U, Wong J, Wong DT, Chung F. Preoxygenation and intraoperative ventilation strategies in obese patients: a comprehensive review. Curr Opin Anaesthesiol. 2016 Feb;29(1):109-18. doi: 10.1097/ACO.0000000000000267. PMID 26545146
- [Background] Jense HG, Dubin SA, Silverstein PI, O'Leary-Escolas U. Effect of obesity on safe duration of apnea in anesthetized humans. Anesth Analg. 1991 Jan;72(1):89-93. doi: 10.1213/00000539-199101000-00016. PMID 1984382
- [Background] Bodily JB, Webb HR, Weiss SJ, Braude DA. Incidence and Duration of Continuously Measured Oxygen Desaturation During Emergency Department Intubation. Ann Emerg Med. 2016 Mar;67(3):389-95. doi: 10.1016/j.annemergmed.2015.06.006. Epub 2015 Jul 9. PMID 26164643
- [Background] Applegate RL 2nd, Dorotta IL, Wells B, Juma D, Applegate PM. The Relationship Between Oxygen Reserve Index and Arterial Partial Pressure of Oxygen During Surgery. Anesth Analg. 2016 Sep;123(3):626-33. doi: 10.1213/ANE.0000000000001262. PMID 27007078
- [Background] Szmuk P, Steiner JW, Olomu PN, Ploski RP, Sessler DI, Ezri T. Oxygen Reserve Index: A Novel Noninvasive Measure of Oxygen Reserve--A Pilot Study. Anesthesiology. 2016 Apr;124(4):779-84. doi: 10.1097/ALN.0000000000001009. PMID 26978143
- [Derived] Tsymbal E, Ayala S, Singh A, Applegate RL 2nd, Fleming NW. Study of early warning for desaturation provided by Oxygen Reserve Index in obese patients. J Clin Monit Comput. 2021 Aug;35(4):749-756. doi: 10.1007/s10877-020-00531-w. Epub 2020 May 18. PMID 32424516

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rainbow Sensor
Started | 80
Completed | 77
Not Completed | 3
Not completed — Equipment Issues | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rainbow Sensor
Number analyzed (Participants) | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 53
  >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 77

OUTCOME MEASURES:

1. Primary Outcome: Utility of ORi Providing Added Warning Time
Description: Evaluate the clinical utility of the change in the oxygen reserve index as an early warning of impending arterial oxygen desaturation in Obese patients (30 < BMI < 40 kg m-2) and Normal BMI patients (19 < BMI < 25 kg m-2).
Time Frame: 1 year
Population: In 4 subjects, the device failed initial calibration. In another subject, clinical care constraints precluded completion of the data collection.
Measure: Number; unit: seconds
Arm/Group | Rainbow Sensor
Number analyzed (Participants) | 72
seconds
  Added warning time in Obese: number analyzed (Participants) | 36
  Added warning time in Obese | 46.5
  Added warning time in Normal BMI: number analyzed (Participants) | 36
  Added warning time in Normal BMI | 87.0

ADVERSE EVENTS:
Time Frame: Approximately 8 hours.
Arm/Group | Rainbow Sensor
All-Cause Mortality (participants affected / at risk) | 0/77
Serious Adverse Events (participants affected / at risk) | 0/77
Other Adverse Events (participants affected / at risk) | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT03021551/Prot_SAP_000.pdf